CLINICAL TRIAL: NCT02176174
Title: Ethnicity and Incidence of Twelve Cardiovascular Diseases: A CALIBER Study
Brief Title: Ethnicity and Onset of Cardiovascular Disease: A CALIBER Study
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Wellcome Trust (Other); National Institute for Health Research, United Kingdom (Other Government); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Julie George, Honorary Research Associate, University College, London
Other Study IDs: CALIBER 13-14; 086091/Z/08/Z (Other Grant/Funding Number: Wellcome Trust); RP-PG-0407-10314 (Other Grant/Funding Number: National Institute for Health Research)
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Abdominal Aortic Aneurysm; Coronary Heart Disease; Sudden Cardiac Death; Intracerebral Haemorrhage; Heart Failure; Ischemic Stroke; Myocardial Infarction; Stroke; Peripheral Arterial Disease; Stable Angina Pectoris; Subarachnoid Haemorrhage; Transient Ischemic Attack; Unstable Angina; Cardiac Arrest
Keywords: Ethnic group; Cardiovascular disease; Atherosclerosis
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Coronary Disease; Death, Sudden, Cardiac; Cerebral Hemorrhage; Heart Failure; Ischemic Stroke; Myocardial Infarction; Stroke; Peripheral Arterial Disease; Angina, Stable; Subarachnoid Hemorrhage; Ischemic Attack, Transient; Angina, Unstable; Heart Arrest; Cardiovascular Diseases; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- White: Self-reported ethnic group of Black, using the United Kingdom Census categories, as recorded in electronic health records.
- Black: Self-reported ethnic group of Black, using the United Kingdom Census categories, as recorded in electronic health records.
- South Asian: Self-reported ethnic group of South Asian, using the United Kingdom Census categories, as recorded in electronic health records.
- Mixed/Other: Self-reported ethnic group of Mixed or other, using the United Kingdom Census categories, as recorded in electronic health records.

SUMMARY:
Specific cardiovascular diseases, such as stroke and heart attack, have been shown to vary by ethnic group. However, less is known about differences between ethnic groups and a wider range of cardiovascular diseases. This study will examine differences between ethnic groups (White, Black, South Asian and Mixed/Other) and first lifetime presentation of twelve different cardiovascular diseases. This information may help to predict the onset of cardiovascular diseases and inform disease prevention strategies.

The hypothesis is that different ethnic groups have differing associations with the range of cardiovascular diseases studied.

DETAILED DESCRIPTION:
There is evidence from epidemiological studies that different ethnic groups are associated with increased incidence of specific cardiovascular diseases. However, the majority of existing studies have examined associations with one or two acute conditions such as stroke or coronary heart disease or focused on a particular ethnic group.

The aim of this study is to examine the differing associations between four ethnic groups and the initial lifetime presentation of a broad range of cardiovascular diseases, including chronic presentations such as stable angina. The hypothesis is that there will be heterogeneity of associations between the different ethnic groups and the full range of cardiovascular diseases studied.

The study will use data from the CALIBER data set of clinically collected electronic health record data from England.

This study is part of the CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records) programme funded over 5 years from the National Institute for Health Research (NIHR) and Wellcome Trust. The central theme of the CALIBER research is linkage of the Myocardial Ischaemia National Audit Project (MINAP) with primary care (Clinical Practice Research Datalink - CPRD) and other resources. The overarching aim of CALIBER is to better understand the aetiology and prognosis of specific coronary phenotypes across a range of causal domains, particularly where electronic records provide a contribution beyond traditional studies. CALIBER has received both Ethics approval (ref 09/H0810/16) and ECC approval (ref ECC 2-06(b)/2009 CALIBER data set).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30 and over
* Registered with a participating general practice during the study period
* Minimum one year of records prior to study entry meeting CPRD data quality

Exclusion Criteria:

* Patients without a record of ethnic group
* Patients without record of gender
* Patients with prior atherosclerotic disease, as recorded in primary care or hospitalisation data
* Pregnant women in the 6 months before the eligibility date

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in the CALIBER database who have a record of ethnic group while registered at one of 225 general practices contributing data to CPRD (the Clinical Practice Research Datalink) and consenting to data linkage.
Sampling Method: Non-Probability Sample
Enrollment: 1068318 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Initial presentation of cardiovascular disease | 10 years
  First recorded diagnosis of cardiovascular disease during follow-up: ventricular arrhythmia / sudden cardiac death, heart failure, unheralded coronary death, myocardial infarction, unstable angina, stable angina, abdominal aortic aneurysm, peripheral arterial disease, subarachnoid haemorrhage, intracerebral haemorrhage, ischaemic stroke, transient ischaemic attack

SECONDARY OUTCOMES:
All cause mortality | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Julie George, Phd, Principal Investigator — University College, London; Harry Hemingway, PhD, Study Director — University College, London

REFERENCES:
- [Background] Denaxas SC, George J, Herrett E, Shah AD, Kalra D, Hingorani AD, Kivimaki M, Timmis AD, Smeeth L, Hemingway H. Data resource profile: cardiovascular disease research using linked bespoke studies and electronic health records (CALIBER). Int J Epidemiol. 2012 Dec;41(6):1625-38. doi: 10.1093/ije/dys188. Epub 2012 Dec 5. PMID 23220717
- [Derived] George J, Mathur R, Shah AD, Pujades-Rodriguez M, Denaxas S, Smeeth L, Timmis A, Hemingway H. Ethnicity and the first diagnosis of a wide range of cardiovascular diseases: Associations in a linked electronic health record cohort of 1 million patients. PLoS One. 2017 Jun 9;12(6):e0178945. doi: 10.1371/journal.pone.0178945. eCollection 2017. PMID 28598987
- See also: CALIBER web site and data portal — https://www.caliberresearch.org/